CLINICAL TRIAL: NCT02804581
Title: Potential Role of Gum Arabic as Immunomodulator In Sudanese Rheumatoid Arthritis Patients
Brief Title: Gum Arabic as Immunomodulator In Rheumatoid Arthritis Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lamis Kaddam (Other)
Collaborators: University of Khartoum (Other); Military hospital (Unknown)
Responsible Party: Sponsor-Investigator, Lamis Kaddam, Dr, Al-Neelain University
Organization: Al-Neelain University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: University of Khartoum
Record Dates: First submitted 2016-06-15; First posted 2016-06-17 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Gum Arabic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gum Arabic (Experimental): Oral intake of 30 gram of Gum Arabic daily for 12 weeks
  Interventions: Dietary Supplement: Gum Arabic

INTERVENTIONS:
Dietary Supplement: Gum Arabic — Oral intake of GA in powder from30 grams per day

SUMMARY:
Gum Arabic (GA) rich dietary fiber it is a water-soluble dietary fiber derived from the dried gummy exudates of the stems and branches of Acacia senegal, GA found to have strong immuno modulator in vitro where it increased IL10 production showing strong anti-inflammatory effects (19).

The aim of this study is to determine the role of gum Arabic in immunomodulation among patients with rheumatoid arthritis.

DETAILED DESCRIPTION:
Butyrate is short chain fatty acids representing the most important end product of colonic bacterial aerobic fermentation of Gum Arabic , it has a potent anti-inflammatory effect and can down regulates TNF a expression by modulating NF-kB-DNA binding activity , in addition butyrate is known to act as histone deacetylase inhibitor in the cells.Recently, in vitro and in vivo data indicates that HDAC inhibitors may have anti-inflammatory effect due to their effects on cell death acting through acetylation of non-histone proteins. The possible anti-rheumatic mechanisms of HDAC inhibitors, including growth arrest in rheumatoid arthritis synovial fibroblasts (RASFs), suppression of pro-inflammatory cytokines, suppressing angiogenesis as well as the protective effects on bone and cartilage against their destruction.

The investigators expect regular intake of GA will raise serum butyrate level. The endogenous butyrate decreases the TNF level. The latter will decrease the number of relapsing episodes, arresting the destruction of joints and improve both survival and life quality of rheumatoid arthritis patients.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of Rheumatoid Arthritis
2. Clinically stable as evidenced by medical history, complete physical examination
3. All medications and dosages are stable for 6 weeks before study entry,
4. Non Pregnant ladies.

Exclusion Criteria:

* 1- hepatic, cardiovascular, pulmonary, malignant, hematologic, neurologic, infectious, or inflammatory diseases unrelated to Rheumatoid arthritis.

  2-Hospital admission within 4 weeks of start of the study.

  3- Uncontrolled hypertension 4- Asthma or severe atopic disease;

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2016-06; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
The level of C reactive protein (CRP)and Tumer necrosis factor alpha TNF | 12 weeks

SECONDARY OUTCOMES:
clinical improvement | 12 weeks
Total anti-oxidant capacity (TAC), malondialdehyde (MDA) and hydrogen peroxide (H2O2) level | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alnour Alagib, MBBS,MD,MRCP, Study Chair — Military hospital; Amal M Saeed, MBBS,PhD, Study Director — University of Khartoum
Locations (1):
- Military Hospital Rheumatology, Khartoum, Umdorman, Sudan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xuan NT, Shumilina E, Nasir O, Bobbala D, Gotz F, Lang F. Stimulation of mouse dendritic cells by Gum Arabic. Cell Physiol Biochem. 2010;25(6):641-8. doi: 10.1159/000315083. Epub 2010 May 18. PMID 20511709
- [Background] Adcock IM. HDAC inhibitors as anti-inflammatory agents. Br J Pharmacol. 2007 Apr;150(7):829-31. doi: 10.1038/sj.bjp.0707166. Epub 2007 Feb 26. PMID 17325655
- [Derived] Kamal E, Kaddam LA, Dahawi M, Osman M, Salih MA, Alagib A, Saeed A. Gum Arabic Fibers Decreased Inflammatory Markers and Disease Severity Score among Rheumatoid Arthritis Patients, Phase II Trial. Int J Rheumatol. 2018 Jul 5;2018:4197537. doi: 10.1155/2018/4197537. eCollection 2018. PMID 30112005